CLINICAL TRIAL: NCT01491529
Title: 13-week, Double-blind, Placebo-controlled, Fixed-dose, Multicenter Study to Evaluate the Efficacy and Safety of Modified Release AFQ056 in Reducing Moderate to Severe L-dopa Induced Dyskinesias in Patients With Parkinson's Disease
Brief Title: Evaluation of the Efficacy and Safety of Modified Release AFQ056 in Parkinson's Patients With L-dopa Induced Dyskinesias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAFQ056A2223; 2011-002074-23 (EudraCT Number)
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2016-03

CONDITIONS: Dyskinesias; Parkinson Disease; Movement Disorders; Parkinsonian Disorders; Anti-Dyskinesia Agents
Keywords: Parkinson Disease; L-dopa; Levodopa; Dyskinesia; Amantadine
MeSH Terms: conditions — Dyskinesias; Parkinson Disease; Movement Disorders; Parkinsonian Disorders | interventions — mavoglurant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- AFQ056 150 mg (Experimental): Patients randomized to the AFQ056 150 mg arm will receive AFQ056 oral tablets to be titrated until reaching the target dose of 150 mg twice daily.
  Interventions: Drug: AFQ056
- AFQ056 200 mg (Experimental): Patients randomized to the AFQ056 200 mg arm will receive AFQ056 oral tablets to be titrated until reaching the target dose of 200 mg twice daily.
  Patients will be randomized in two groups by amantadine status.
  * Group 1: Patients are not permitted to take amantadine within 2 weeks prior to the BL1 visit.
  * Group 2: Patients must be on a stable and well tolerated dose of amantadine for at least 4 weeks prior to BL1 and must maintain the stable dose of amantadine during the remainder of the study.)
  Interventions: Drug: AFQ056
- Placebo (Placebo Comparator): Patients randomized to the Placebo arm will receive oral AFQ056 Placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AFQ056 — AFQ056 will be supplied as oral modified release tablets in 25 mg, 50 mg, 100 mg, 150 mg, and 200 mg.
  Patients will be randomized in two groups by amantadine status.
  * Group 1: Patients are not permitted to take amantadine within 2 weeks prior to the BL1 visit.
  * Group 2: Patients must be on a stable and well tolerated dose of amantadine for at least 4 weeks prior to BL1 and must maintain the stable dose of amantadine during the remainder of the study.)
  Arms: AFQ056 150 mg; AFQ056 200 mg
Drug: Placebo — Placebo for AFQ056 will be supplied as oral tablets.
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety of modified release AFQ056 in patients that have Parkinson's Disease L-dopa Induced Dyskinesias (PD-LID)

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 30-80 years old
* Use of highly effective methods of contraception during study in women of childbearing potential
* Outpatients
* Clinical diagnosis of Parkinson's Disease according to UK Parkinson's Disease Society Brain Bank Clinical Diagnosis criteria
* Score of >/= 2 on UPDRS items 32 and 33
* Dyskinesias for at least 3 months before baseline
* On stable treatment regimen with L-dopa and other anti-parkinsonian treatment for 4 weeks prior to baseline
* Demonstrate capacity to complete accurate diary ratings
* Patients who have a primary caregiver willing to assess the condition of the patient throughout the study in accordance with protocol requirements
* Group 2 only: Patients must be on a stable and well tolerated dose of amantadine for at least 4 weeks prior to BL1 and must maintain the stable dose of amantadine during the remainder of the study

Exclusion Criteria:

* Atypical/secondary form of Parkinson's disease
* History of surgical treatment of PD, including deep brain stimulation
* A score of 5 in the "ON"- state on the Modified Hoehn and Yahr scale
* Advanced, severe, or unstable disease other than PD
* Evidence of dementia
* Treatment with certain prohibited medications
* Amantadine within 2 weeks prior to BL1 visit (applies to Group 1 only)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in modified AIMS (Abnormal Involuntary Movement Scale) total score from baseline to Week 12 | 12 weeks
  The modified AIMS is a scale used to assess dyskinesia. It focuses on six different parts of the body and rates abnormal movements from 0 (absence of dyskinesia to 4 (severe) (maximal score, 24).
  Change from baseline to Week 12 will be analyzed using the mixed effect repeated measures model (MMRM) including treatment, pooled center, week, treatment by week interaction as fixed effects and baseline total score as covariate with an unstructured covariance structure.
The incidence rate of adverse events | Monitored for the duration of the study which is 13 weeks
  The occurrence of adverse events would be sought by non-directive questioning of the patient. Adverse events may also be detected when they are volunteered by the patient or through physical examination, laboratory test, or other assessments.
  AEs will be summarized by presenting, for each treatment group the number and percentage of patients having any adverse event, having an adverse event in each system organ class and having each individual adverse event by system organ class and preferred term.
Time to onset of adverse events | Monitored for the duration of the study which is 13 weeks
  The occurrence of adverse events (AEs) would be sought by non-directive questioning of the patient. Adverse events may also be detected when they are volunteered by the patient or through physical examination, laboratory test, or other assessments.
  AEs will be summarized by presenting, for each treatment group the number and percentage of patients having any adverse event, having an adverse event in each system organ class and having each individual adverse event by system organ class and preferred term.
The percentage of patients reaching and maintaining the target dose during the fixed dose treatment period | Assessed during the fixed dose treatment period of 6 weeks
  Randomized patients will be up titrated to the target dose and remain on the target dose for the duration of the fixed dose treatment period.
  AEs will be summarized by presenting, for each treatment group the number and percentage of patients having any adverse event, having an adverse event in each system organ class and having each individual adverse event by system organ class and preferred term.
The percentage of patients discontinued during the up titration period due to AE | Assessed during the up titration period of 6 weeks
  Patients randomized will be up titrated to the target doses at regular intervals during the up titration period.
  AEs will be summarized by presenting, for each treatment group the number and percentage of patients having any adverse event, having an adverse event in each system organ class and having each individual adverse event by system organ class and preferred term.

SECONDARY OUTCOMES:
The change in total score and sub-score of UDysRS Parts I, II, III, and IV from baseline to Week 12 | 12 weeks
  The UDysRS captures dyskinesia and has 4 parts: I: Historical Disability of On-Dyskinesia impact (max 44 pts); II: Historical Disability of Off-Dystonia impact (max 16 pts); III: Objective Impairment dyskinesia (max 28 pts); IV: Objective Disability based on Part III activities (max 16 pts). Higher scores mean greater severity.
  Change from baseline to Week 12 will be analyzed using mixed-effect repeated measure model (MMRM) including treatment, pooled center, week, treatment by week interaction as fixed effects and baseline total score as covariate with an unstructured covariance structure.
Change in Lang-Fahn Activities of Daily Living Dyskinesia Scale (LFADLDS) total score from baseline to Week 12 | 12 weeks
  The LFADLDS assesses the degree of dyskinesia interfering with activities of daily living. Specific definitions for severity rating codes (range, 0-4 for each task) will be provided for reproducibility of results. A higher score indicates more severe impairment. A patient and caregiver version of the revised LFADLDS will be used in this study.
  Change from baseline to Week 12 will be analyzed using MMRM including treatment, pooled center, week, treatment by week interaction as fixed effects and baseline total score as covariate with an unstructured covariance structure.
Change in clinician-rated global impression of change (CGIC) score from baseline to Week 12 | 12 weeks
  The CGIC provides investigator-rated assessment of change from baseline to assess disability due to dyskinesia. Change from baseline will be rated on a 7-point, Likert-type scale where 1 = markedly improved, 2 = moderately improved, 3 = minimally improved, 4 = unchanged, 5 = minimally worse, 6 = moderately worse, and 7 = markedly worse.
  The CGIC score at week 12 last observation carried forward (LOCF) will be analyzed using analysis of covariance (ANCOVA) model with treatment group, pooled center, and baseline CGIS (Clinical Global Impression of Severity) score as factors.
Change from baseline Total ON- and OFF-times and ON-time with dyskinesia and with troublesome dyskinesias (patient diary) to Week 12 | 12 weeks
  A patient home diary developed and validated for use in PD patients will be used to record whether the patient is asleep, OFF, ON without dyskinesia, ON with troublesome dyskinesias, and ON with non-troublesome dyskinesia.
  Change from baseline to Week 12 will be analyzed using MMRM including treatment, pooled center, week, treatment by week interaction as fixed effects and baseline total score as covariate with an unstructured covariance structure.
Change in score for items 32, 33 and 34 of Part IV of the Unified Parkinson's Disease Rating Scale (UPDRS ) from baseline to Week 12 | 12 weeks
  UPDRS assesses the disease state of PD. Question 32 assesses length of dyskinesias in percentage of the day. Question 33 assesses disability during the previous week (not disabling, mildly disabling, moderately disabling, severely disabling, completely disabling). Question 34 assesses painfulness of dyskinesias from 0 (no painful dyskinesias) to 4 (marked).
  The change will be analyzed using MMRM including treatment, pooled center, week, treatment by week interaction as fixed effects and baseline total score as covariate with an unstructured covariance structure.
Changes in vital signs from baseline to each post-baseline visit | Monitored at regular visits throughout duration of the study which is 13 weeks
  Pulse and blood pressures are taken at each visit. Vital sign data will be summarized by presenting summary statistics for change from baseline values. The incidence rates of clinically notable vital sign abnormalities will be summarized.
Changes in hematology/blood chemistry and urinalysis laboratory evaluations from baseline to each post-baseline visit where hematology/blood chemistry and urinalysis are collected | Monitored at regular visits throughout duration of the study which is 13 weeks
  Standard hematology with differential; measures of coagulability: aPTT, PT/INR; standard clinical chemistry; FSH, LH, oxytocin, prolactin, TBG, TSH, and T4; urinalysis (specific gravity, protein, glucose and blood) Laboratory data will be summarized by presenting shift tables, by presenting summary statistics, change from baseline values, and incidence rates of clinically notable abnormalities summarized.
Changes in electrocardiogram (ECG) from baseline to each post-baseline visit where ECGs are performed | Monitored at regular visits throughout duration of the study which is 13 weeks
  A standard 12-lead ECG will be performed. A central facility will be used for interpretation and analysis of the ECGs.
  ECG intervals will be summarized by summary statistics for change from baseline values and incidence rates of clinically notable abnormalities summarized.
Percentage of adverse events including treatment emergent adverse events and serious adverse events | Monitored for the duration of the study which is 13 weeks
  The occurrence of adverse events would be sought by non-directive questioning of the patient. Adverse events may be detected when they are volunteered by the patient or through physical examination, laboratory test, or other assessments.
  Treatment-emergent adverse events (TEAEs) will be summarized by presenting, for each treatment group, the number and percentage of patients having an AE, having an AE in each system organ class and having each AE by system organ class and preferred term.
Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part III (Motor Examination) scores from baseline to Week 12 | 12 weeks
  Part III of the UPDRS (items 18-31; score 0-56), measures speech, facial expression, tremor, action or postural tremor, rigidity, finger taps, hand movement, alternating movement, leg agility, arising from a chair, posture, gait, postural stability, and bradykinesia. A higher score means worsening of symptoms.
  Changes from baseline to Week 12 will be analyzed using MMRM including treatment, pooled center, week, treatment by week interaction as fixed effects and baseline total score as covariate with an unstructured covariance structure.
Change in Mini Mental State Exam (MMSE) total scores from baseline to Week 12 | 12 weeks
  The MMSE is a test of cognitive dysfunction consisting of orientation, registration, attention-calculation, recall, and language administered by a health care professional. The MMSE results in total possible score of 30, with higher scores meaning better function.
  The change from baseline to endpoint at Week 12 in MMSE total score will be analyzed using LOCF ANCOVA with treatment group and pooled center as factors and the baseline score as a covariate. Treatment differences in the change from baseline for scores with 90% CI will be reported as descriptive statistics.
Change in cognitive test battery (CogState) scores form baseline to Week 12 | 12 weeks
  This test consists of: Detection Task, Identification Task, One Card Learning Task, One Back Task, and International Shopping List Task. Speed times and working memory will be measured by the number of correct responses.
  The change from baseline to endpoint at Week 12 for cognitive function will be analyzed using LOCF ANCOVA with treatment group and pooled center as factors and the baseline score as a covariate. Treatment differences in the change from baseline for cognitive function with 90% CI will be reported as descriptive statistics
Total scores of the Scales for Outcomes in Parkinson's disease - Psychiatric Complications (SCOPA-PC) | Assessed for 12 weeks
  The SCOPA-PC is an easily administered semi-structured, questionnaire developed for the assessment of psychiatric symptoms in Parkinson's disease patients administered by a clinician with input provided by patient and caregiver. The total SCOPA score ranges from 0-21, with higher scores reflecting more psychiatric complications.
  The SCOPA-PC total score and each of the item scores will be summarized.
Proportion of patients who have suicidal ideation and behavior as mapped to Columbia Classification Algorithm for Suicide assessment (C-CASA) using data from Columbia-Suicide Severity Rating Scale (C-SSRS) | This will be assessed for the duration of the study which is 13 weeks
  The C-SSRS assesses suicidal ideation/behavior using a patient interview. The data is mapped to Columbia Classification Algorithm for Suicide assessment. The code and categories are: completed suicide, suicide attempt, preparatory actions toward imminent suicide behavior, suicidal ideation, self-injurious behavior without suicidal intent.
  The proportion of patients who are coded in the categories above, the proportion of patients with any suicidal behavior engaged in during the study, and the proportion of patients with suicidality will be summarized.
Plasma Pharmacokinetics of AFQ056 in patients with Parkinson's disease with moderate to severe dyskinesias | At Week 12 or earlier if the patient discontinues the study before Week 12
  Blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein. The first blood sample will be collected 1-3 hours after morning study medication dose. The second sample will be collected 3-5 hours after the morning study medication dose. The third blood sample will be collected 5-7 hours after the morning study medication dose.
  Summary statistics for concentrations per sampling window will be provided and average plasma levels will be calculated.
Pharmacokinetics of AFQ056 in patients with Parkinson's disease with moderate to severe dyskinesias | Monitored at regular visits throughout duration of the study which is 13 weeks
  Blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein. An alternative sampling method will also be explored. At all visits, the sample will be collected 1-3 hours after morning study medication dose. At Week 12, the second sample will be collected 3-5 hours after the morning study medication dose and the third sample will be collected 5-7 hours after the morning study medication dose.
  Summary statistics for concentrations per sampling window will be provided and average plasma levels will be calculated.
Investigate the safety of concomitant administration of AFQ056 with amantadine | 12 weeks
  Investigation of the safety of AFQ056 with concomitant amantadine is being studied to gather drug-drug interaction data of amantadine and AFQ056 in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- United States (5):
  - Novartis Investigative Site, Sunnyvale, California
  - Novartis Investigative Site, Englewood, Colorado
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Austria (3):
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, London, Ontario, Canada
- France (4):
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Poitiers
- Germany (8):
  - Novartis Investigative Site, Beelitz-Heilstätten
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Stadtroda
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Szeged
- Italy (4):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Bolzano, BZ
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Bratislava, Slovakia
- Spain (4):
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne

REFERENCES:
- [Derived] Trenkwalder C, Stocchi F, Poewe W, Dronamraju N, Kenney C, Shah A, von Raison F, Graf A. Mavoglurant in Parkinson's patients with l-Dopa-induced dyskinesias: Two randomized phase 2 studies. Mov Disord. 2016 Jul;31(7):1054-8. doi: 10.1002/mds.26585. Epub 2016 May 23. PMID 27214258
- See also: Results for CAFQ056A2223 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=11843